CLINICAL TRIAL: NCT01430598
Title: Randomized Single Blinded Study Comparing Patient Function and Satisfaction With Arthroscopic Subacromial Decompression Before and After Repair of Complete Rotator Cuff Tears
Brief Title: Study Comparing Patient Function and Satisfaction With Arthroscopic Subacromial Decompression Before and After Repair of Complete Rotator Cuff Tears
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Lauren Suchy, Academic Research Coordinator, Ascension Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ME 11 0021
Record Dates: First submitted 2011-08-29; First posted 2011-09-08 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Rotator Cuff Tear; Acromial Spur
Keywords: Full Thickness Rotator Cuff Tear and Acromial Spur
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Subacromial decompression before repair of a complete rotator cuff tear.
  Interventions: Procedure: Rotator Cuff Repair and Subacromial Decompression; Other: Questionnaire
- B (Active Comparator): Subacromial decompression after repair of a complete rotator cuff repair.
  Interventions: Procedure: Rotator Cuff Repair and Subacromial Decompression; Other: Questionnaire

INTERVENTIONS:
Procedure: Rotator Cuff Repair and Subacromial Decompression — Arthroscopic decompression and rotator cuff repair will be completed during the same surgical date.
Other: Questionnaire — Patients will be asked to complete two separate questionnaires prior to the surgical intervention. Patients will be asked to complete the same two questionnaires at 12 weeks post surgery.

SUMMARY:
The investigators aim to establish whether completing a subacromial decompression before or after repair of a complete rotator cuff tear has any clinical significance. Both the arthroscopic decompression and rotator cuff repair will be completed during the same surgical date. The investigators null hypothesis contends that full-thickness rotator cuff tear repair performed before versus after subacromial decompression will not influence patient's post-operative pain or functionality.

DETAILED DESCRIPTION:
All patients with a diagnosed full thickness rotator cuff tear and symptomatic subacromial decompression will be consulted about arthroscopic subacromial decompression and rotator cuff repair. The possible risks and benefits will be discussed with the patient in detail by the operating surgeon. If a patient agrees to undergo surgical intervention (i.e. arthroscopic subacromial decompression and rotator cuff repair in the same surgical setting), they will be approached and informed regarding involvement in the study. This is a single blind study so participants will not know into which arm they have been randomized.

Once consented, the subject will be randomized into one of two treatment arms. Those in Arm A will have subacromial decompression before repair of a complete rotator cuff and those in Arm B will have subacromial decompression after repair of a complete rotator cuff.

Prior to surgical intervention all patients will complete two separate questionnaires in the waiting room. The results of the questionnaires will be later used to compare pre-operative and post-operative changes following shoulder surgery.

On the date of surgery, the operative surgeon will ensure a full-thickness rotator cuff tear is present with an associated acromial spur. If both are present, the operative surgeon will perform the surgical intervention in the previously assigned order according to the patient's treatment arm. All acromial spurs will be burred to a level flush with the remaining non-pathologic acromion. The full-thickness rotator cuff will be repaired utilizing sutures and suture anchors. The specific pattern of repair will be determined intra-operatively. This is standard procedure for arthroscopic rotator cuff repair and subacromial decompression. There is no known risks within the orthopedic literature with performing subacromial decompression before versus after rotator cuff repair. As such, this study aims to identify any significance of the order of surgery if it exists.

Post-operatively all patients will be placed within a Berg SlingShot®. All patients will undergo a period of immobilization within the sling. Patients will be evaluated at 2 weeks, 6 weeks, and 12 weeks post-operatively. The shoulder range of motion and relative strength, compared to the contralateral limb, will be assessed. They will be prescribed formal physical therapy in the outpatient setting. At the 12 week visit each subject will complete the questionnaires once again. The scores will be tabulated and inserted in the Excel spreadsheet.

The pre-operative and post-operative scores will be compared. The change in score from each treatment arm will be averaged and analyzed for statistically significant difference. Also, the pre- and post-operative forward flexion, abduction range of motion will be compared. The external and internal rotation strengths will be compared from the pre- and post-operative evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* Symptomatic patients with MRI positive full thickness rotator cuff tears
* Clinically and/or radiographically positive subacromial impingement/spur with associated rotator cuff tendonitis and bursitis
* Patients who have failed outpatient conservative therapy, including, but not limited to physical therapy and subacromial injection with steroid and local anesthetic

Exclusion Criteria:

* Patient with radiographic evidence of glenohumeral degenerative joint disease or rotator cuff arthropathy
* Patients with a prior history of joint sepsis
* Patients who have had previous shoulder surgery on the anticipated operative limb
* Patients with a diagnosed pathology causing associated pain and/or weakness to the anticipated operative limb
* Patient deemed unable to complete the post-operative rehabilitation protocol
* Patients diagnosed, either intra-operatively or by MRI, as having irreparable rotator cuff tears

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Pre and Post Surgery Pain and Satisfaction | 1 year
  Both arms will complete an identical baseline and post-operative pain and functionality survey. The data will be analyzed to determine the rate of change between the pre and post surgery results. The results from the two groups will be compared to determine if there is a significant difference in pain and functionality between subjects in Arm A and Arm B.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Genesys Regional Medical Center-General Surgery Center, Grand Blanc, Michigan
  - Greater Flint Sports Medicine, Grand Blanc, Michigan